CLINICAL TRIAL: NCT06397872
Title: A Phase 1, Multi-center, Open-label Study to Evaluate the Pharmacokinetics, Safety, and Tolerability of Multiple Oral Doses (6 Days) of 100 mg Resmetirom in Subjects With Severe Renal Impairment and in Matched Healthy Control Subjects With Normal Renal Function
Brief Title: A Study to Evaluate the Pharmacokinetics, Safety, and Tolerability of Multiple Oral Doses (6 Days) of 100 mg Resmetirom in Subjects With Severe Renal Impairment and in Matched Healthy Control Subjects With Normal Renal Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Madrigal Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MGL-3196-21
Record Dates: First submitted 2024-04-30; First posted 2024-05-03 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Renal Impairment
MeSH Terms: conditions — Renal Insufficiency | interventions — resmetirom

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Severe renal impairment (Experimental)
  Interventions: Drug: 100 mg Resmetirom Tablet
- Normal Healthy Match (Experimental): Matched to severe renal impairment
  Interventions: Drug: 100 mg Resmetirom Tablet

INTERVENTIONS:
Drug: 100 mg Resmetirom Tablet — Once daily oral dose for 6 days
  Other Names: Rezdiffra, MGL-3196

SUMMARY:
The purpose of this study is to directly characterize the pharmacokinetic (PK) profiles of resmetirom and its major metabolite (MGL-3623) following oral administration of 100 mg resmetirom (QD x 6 days) in subjects with severe renal impairment (RI) compared to healthy matched control subjects with normal renal function.

ELIGIBILITY:
Inclusion Criteria:

* Capable of understanding the informed consent and willing and able to provide written informed consent.

Subjects with Severe Renal Impairment

* Body weight > 50 kg, BMI between 18.0 to 45.0 kg/m2, inclusive, at the screening visit.
* Impaired renal function with estimated glomerular filtration rate (eGFR) < 30 mL/min/1.73 m2, determined using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) creatinine equation at the screening visit and not requiring dialysis.
* Stable renal function with no clinically significant change in renal status at least 29 days prior to first dosing and is not currently or has not been previously on dialysis for at least 1 year.
* With exception of the known renal disease and stable comorbidities, is in otherwise good health, in the opinion of the Investigator, based on medical history, physical examination, vital sign measurements, ECG, and clinical laboratory tests performed at the screening and Day -1 visits.

Matched Healthy Control Subjects

* Must match the BMI (within ± 20%) of a subject with severe RI.
* Must match the age (± 10 years) and sex of a subject with severe RI.
* Normal renal function with eGFR ≥ 90 mL/min/1.73 m2, determined using the CKD-EPI creatinine equation (2021) at the screening and Day -1 visit.
* Must be in good health as determined by medical history, physical examination, vital sign measurements, ECG, and clinical laboratory tests at the screening and Day -1 visits.

Exclusion Criteria:

All Subjects

* Gilbert's syndrome.
* Pre-existing condition interfering with normal gastrointestinal anatomy or motility, or hepatic function that could interfere with the absorption, metabolism, and/or excretion of study drug (cholecystectomy is allowed).

Subjects with Severe Renal Impairment

* TSH < 0.3 or > 7 mIU/L at the screening or Day -1 visit.
* Evidence or history of clinically significant hematological, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, neurological, or psychiatric disease, except for stable comorbidities.
* Has had a failed renal transplant or has had a nephrectomy.
* Has end stage renal disease requiring dialysis.
* Systolic blood pressure outside the range of 80 to 170 mmHg, diastolic blood pressure outside the range of 40 to 100 mmHg, or heart rate outside the range of 40 to 100 bpm at the screening or Day -1 visit.

Healthy Matched Control Subjects

* Current or recent (< 6 months from the screening visit) hepatobiliary disease; or serum aspartate aminotransferase (AST), alanine aminotransferase (ALT), or direct bilirubin value greater than the upper limit of reference range at the screening or Day -1 visit.
* TSH outside normal range.
* Evidence or history of clinically significant hematological, endocrine, pulmonary, gastrointestinal, cardiovascular, renal, hepatic, neurological, or psychiatric disease.
* Systolic blood pressure outside the range of 90 to 160 mmHg, diastolic blood pressure outside the range of 40 to 95 mmHg, or heart rate outside the range of 40 to 100 bpm at the screening or Day -1 visit.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2024-03-06 (Actual); Primary Completion 2024-09-16 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Plasma pharmacokinetics - Cmax | 8 days
  Cmax after administration
Plasma pharmacokinetics - Tmax | 8 days
  Tmax after administration
Plasma pharmacokinetics - AUC(0-Last) | 8 days
  AUC(0-Last) after administration
Plasma pharmacokinetics - t1/2 | 8 days
  t1/2 after administration

SECONDARY OUTCOMES:
Effect on the incidence of adverse events | 13 days

CONTACTS AND LOCATIONS:
Overall Officials: Geoff Rezvani, Study Director — Madrigal Pharmaceuticals, Inc.
Locations (3):
- United States (3):
  - Madrigal Research Center, Orlando, Florida
  - Madrigal Research Center, Tampa, Florida
  - Madrigal Research Center, Chicago, Illinois